CLINICAL TRIAL: NCT04823351
Title: Randomized Controlled Trial to Compare Clinical Efficacy of Surgical and Filtering Facepiece 2 Masks for Care Home Workers Treating COVID-19 Patients
Brief Title: Clinical Efficiency of Surgical Masks and Filtering Face-piece 2 Masks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); ETH Zurich (Other); Kantonsspital Winterthur KSW (Other); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 4078P0_198258
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The objective is to perform a cluster-randomized, parallel, controlled, non-inferiority study among Swiss nursing and retirement homes to evaluate the efficacy of surgical masks vs. FFP2 masks during patient care and prospectively observe possible infections amongst both vaccinated and unvaccinated staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFP2 Mask (Other): Universal FFP2-masking for every healthcare worker with patient contact, compared to selective FFP2-masking, which means that FFP2 masks are worn only during aerosol-generating procedures such as tube manipulation;
  Interventions: Behavioral: Surgical Mask
- Surgical Mask (Other): Universal surgical mask IIR type masking for healthcare workers in contact with COVID-19 patients.
  Interventions: Behavioral: Surgical Mask

INTERVENTIONS:
Behavioral: Surgical Mask — The randomized wards will be wearing either FFP2 masks or surgical masks for 8 weeks. Then a cross-over will occur for another 8 weeks.

SUMMARY:
Recent results demonstrated an increased risk of COVID-19 infection among healthcare workers (HCW), particularly when access to personal protective equipment (PPE) was inadequate. (ref). During the COVID-19 pandemic, access to PPE has become complicated by a surge in worldwide demand combined with production limitations and logistical barriers. Since their introduction in hospitals in the 1990s, filtering facepiece (FFP) masks, mostly of the FFP2 type, are used by HCWs to protect themselves against bioaerosols due to tuberculosis, measles, and selected respiratory viruses. The COVID-19 pandemic has sparked debate around reasonable and safe use of the different types of face masks to protect the HCWs who provide direct care for COVID-19 patients. At the heart of the discussion are the respective contributions to SARS-CoV-2 transmissions by droplets and aerosols, and the corresponding risk levels resulting in COVID-19 infection.

The objective is to perform a cluster-randomized, parallel, controlled, non-inferiority study among Swiss nursing and retirement homes to evaluate the efficacy of surgical masks vs. FFP2 masks during patient care and prospectively observe possible infections amongst both vaccinated and unvaccinated staff.

Staff in nursing homes will be randomized to use either surgical or FFP2 masks for patient care consistently. Considering an attack rate of 0.8% over three months among healthcare workers, a non-inferiority margin of 5%, and an intracluster variability of 0.01, - we require a minimum of 625 participants per group. The COVID-19 attack rate will be tested by initial serology testing and weekly pooled saliva specimen for SARS-CoV-2 testing. (Re)-Infections will be tracked by weekly pooled saliva-based PCR testing. Exposure to COVID-19 other than during work time will be explored by questionnaires and focus group discussions.

DETAILED DESCRIPTION:
1. Project summary Recent results demonstrated an increased risk of COVID-19 infection among healthcare workers (HCW), particularly when access to personal protective equipment (PPE) was inadequate. (ref) During the COVID-19 pandemic, access to PPE has become complicated by a surge in worldwide demand combined with production limitations and logistical barriers. Since their introduction in hospitals in the 1990s, filtering facepiece (FFP) masks, mostly of the FFP2 type, are used by HCWs to protect themselves against bioaerosols due to tuberculosis, measles, and selected respiratory viruses. The COVID-19 pandemic has sparked debate around reasonable and safe use of the different types of face masks to protect the HCWs who provide direct care for COVID-19 patients. At the heart of the discussion is whether droplets or aerosols transmit SARS-CoV-2, and which of the two is responsible for what risk level of SARS-CoV-2 transmission resulting in disease.

   The objective is to perform a cluster-randomized, parallel, controlled, non-inferiority study among Swiss nursing and retirement homes (homes) to evaluate the efficacy of surgical masks vs. FFP2 masks during patient care and prospectively observe possible infections amongst both vaccinated and unvaccinated staff.

   Staff in nursing homes will be randomized to use either surgical or FFP2 masks for patient care consistently. Considering an attack rate of 0.8%[1] over three months among healthcare workers, a non-inferiority margin of 5%, and an intracluster variability of 0.01,[2] - we require a minimum of 625 participants per group.[3] The COVID-19 attack rate will be tested by initial serology testing and weekly pooled saliva specimen for SARS-CoV-2 testing. (Re)-Infections will be tracked by weekly pooled Saliva based PCR testing. Exposure to COVID-19 other than during work time will be explored by questionnaires and focus group discussions.
2. Study protocol 2.1 State of research in the field 2.1.1 Transmission of COVID-19 by droplets or aerosols Since the beginning of the COVID-19 pandemic, more than 110 million cases were confirmed with almost 2.4 million deaths as of February 22nd, 2020. Given that SARS-CoV-2 is a respiratory virus, its spread is expected to occur mainly by droplets (diameter >5µm) and via contact; however, laboratory tests suggest that SARS-CoV-2 may remain viable and infectious also in aerosols (diameter <5 µm).1,2. Both droplets and aerosols are naturally produced by humans when breathing, talking, coughing, or sneezing. A cough and a sneeze can generate between 3000 and 40,000 droplets of diameters between 0.5 to 12 µm, respectively 3-5; furthermore, droplets and aerosols can both contain SARS-CoV-2 virus if produced by COVID-19 patients. Aerosols are small-size droplets remaining in the air, and thus may travel beyond 2m from a source the respiratory tract bypassing surgical masks. Therefore, healthcare workers have been advised to wear FFP2 masks in procedures that generate aerosols. It remains to be clarified if surgical masks are inferior to FFP2 masks in the care of COVID-19 patients other than being exposed to aerosol-generating procedures. Recent data suggests that if worn correctly by both patient and exposed staff, surgical masks are able of filtering over 90% of particles generated 6.

Specifics about COVID-19 disease transmission and infectious dose are currently lacking. However, numbers in the order of 1000 droplets and more are realistic assumptions.7 The infection risk by one virus copy in viral shedding is about 1.5×10-6 to 1.6×10-5. Thus the infection risk due to aerosols at distances larger than 1-2 meters is substantially lower than that due to close interaction within 1 meter.

Consequently, protection from COVID-19 patients must focus on close interaction where droplets play a significant role, which could be addressed by wearing a surgical mask.

The added protective benefit of FFP2 masks outside so-called "aerosol-generating procedures" where aerosols are believed to be produced in large quantities is meager. Thus, recommending FFP2 masks for non-aerosol-generating procedures with regard to COVID-19 is not justified. Hence, a randomized trial to test the non-inferiority of surgical masks in COVID-19 care (other than during aerosol-generating procedures) is ethically sound.

With logistical challenges arising to vaccinate the greater public8, many people refusing vaccinations, a significant percent of the population having contracted COVID-19 since the beginning of the pandemic, and new mutations emerging with growing amounts of reports of reinfections,9 we are facing a reality in which, regarding their infection and vaccination status, non-homogenous groups of people will have to learn to co-exist for months and possibly years to come.

In Switzerland, there is currently a lot of discordance between hospitals when it comes to the choice of mask for healthcare workers, making recruitment of sufficient participants basically impossible. We decided to focus on including retirement homes and homes for the elderly. The homes have designated wards for COVID-19 and separate wards for patients requiring aerosol generating procedures. They also require more nursing and support staff to take care of the elderly, making them ideal candidates for our study design and tracking infections based on the mask type. In the United States a third of all COVID-19 related deaths in the United States are believed to be linked to nursing homes10, highlighting the importance to have unanimous guidelines as to the most important basic measures such as mask wearing, to reduce infections and mortality across populations.

2.1.2 Face masks and their appropriate use

Two different types of face masks are distinguished for patient care:

Surgical masks (usually II and IIR) have the main role of limiting the transmission of infective agents from HCWs to patients, mainly during surgical procedures. In specific situations such as colonization with multidrug-resistant microorganisms in the respiratory tract or during outbreaks with respiratory pathogens, wearing them is also recommended for infected patients as source control to limit transmission. The fitting of these masks is loose and leakage occurs around the edges of the mask. While IIR masks protect the wearer from projected splashes of biological fluids, they do not provide the wearer with a reliable protection level from inhaling smaller airborne particles unless modified by e.g. knotting the edges. Ref 6

Class 2 filtering facepiece (FFP 2) masks offer respiratory protection for the wearer. They have tight-fitting and minimal leakage occurs around the edges of the mask. Filtering facepiece masks were initially intended to protect workers from dust exposure. However, FFP2 masks were introduced to healthcare predominantly to protect healthcare workers exposed to patients with tuberculosis or measles. (ref) Their appropriate use during the COVID-19 pandemic in healthcare units remains controversial, as explained above. A recent meta-analysis pooling five randomized-controlled trials showed no difference between surgical masks and FFP masks for outcomes such as clinical respiratory illness or laboratory-confirmed influenza. 11 2.2 Aims Primary outcome: The aim of this study is to test the hypothesis that surgical masks are not inferior to FFP2 masks in patient care (in situations outside of aerosol-generating procedures).

Secondary outcome: By including staff who may have received vaccination we want to track possible infections

2.3 Methods

A cluster-randomized, parallel, controlled, non-inferiority study among Swiss nursing- and retirement homes hosting COVID-19 patients will evaluate the benefits of wearing surgical masks vs. FFP2 masks during COVID-19 patient care (outside aerosol-generating procedures).

2.3.1 Settings: Any Swiss nursing- and retirement home offering COVID-19 care is eligible to be included. The homes will be recruited through direct contact. Each home will have an appointed onsite investigator for communication with the study team.

2.3.2 Study duration We will recruit homes between January 1 and March 10th. During three months, the intervention will last until no later than June 30, 2021.

2.3.3.Randomization: Home wards will be computer-randomized before starting the intervention, stratified by ward size.

Intervention: Interventions include either universal FFP2-masking for every healthcare worker with patient contact, compared to selective FFP2-masking, which means that FFP2 masks are worn only during aerosol-generating procedures such as tube manipulation; for all other procedures, healthcare workers wear a surgical mask of the IIR type. Furthermore, weekly saliva-based pooling will be conducted to track possible (re)-infections.

2.3.4 Outcomes: Primary outcomes are new SARS-CoV-2 infections among healthcare workers appointed to deliver care to COVID-19 patients, measured by a baseline seroprevalence testing and a weekly pooled saliva specimen-based SARS-CoV-2 testing. Secondary outcomes are newly identified SARS-CoV-2 infections among healthcare workers by rtPCR; questionnaires on monthly activity for healthcare workers; focus group discussions on workplace vs. private exposure to COVID-19 patients. Serology testing and saliva-based testing for healthcare workers are voluntary and are performed upon written informed consent.

2.3.5 Sample collection and laboratory testing: Sample size calculation: We hypothesize an attack rate of 0.8 % among healthcare workers (0.8% of the participating healthcare workers become SARS-CoV-2 positive by the end of the study period), the surgical masks are non-inferior to FFP2 masks by 5%. Considering an attack rate of 0.8 %, an inferiority margin of 5%, and an intra-cluster correlation coefficient of 0.01, 1250 participants (625 per group) have to be included (one-sided and with 80% power). The study will be conducted in a cross-over design.

2.3.6 Outcome measurements SARS-CoV-2 serology at baseline and weekly saliva-based specimen pooled SARS-CoV-2 tests. Exposure to COVID-19 patients and risk behavior by questionnaire. Qualitative interpretation of focus group discussions.

2.3.7 Data analysis A non-inferiority difference of proportions test will model the primary outcome. Secondary outcomes will be analyzed descriptively.

2.4 Expected Results

We expect that selective FFP2-masking is not inferior to universal FFP-2 masking; however, selecting when and how FFP-2 masks are to be worn by HCWs is not trivial. This project aims to inform those decisions with improvements in our understanding of the issues involved and the generation of on-site data to guide decision-making.

2.5 Project milestones and timeline[15]

2.6 The potential impact of the research Recent research and government regulations6,12 have shown a significant disparity in opinions regarding the appropriate usage of surgical masks / FFP2 masks. In light of new regulations enforcing FFP2 mask usage by the general population in neighboring countries such as Germany and the diverging opinions amongst health care professionals - we expect this study to help elucidate appropriate use and clear up possible misconceptions. Given the lack of research in this area, this study's outcome will potentially have a world-wide public health impact and aid regulatory bodies to make founded decisions and recommendations to both healthcare workers and the public alike.

2.7 Budget (see Excel)

3 References

1. Li P, Fu J-B, Li K-F, et al. Transmission of COVID-19 in the terminal stages of the incubation period: A familial cluster. Int J Infect Dis 2020;96:452-3.
2. van Doremalen N, Bushmaker T, Morris DH, et al. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med 2020;382(16):1564-7.
3. Cole EC, Cook CE. Characterization of infectious aerosols in health care facilities: an aid to effective engineering controls and preventive strategies. Am J Infect Control 1998;26(4):453-64.
4. Wei J, Li Y. Airborne spread of infectious agents in the indoor environment. Am J Infect Control 2016;44(9 Suppl):S102-8.
5. Bourouiba L. Turbulent Gas Clouds and Respiratory Pathogen Emissions: Potential Implications for Reducing Transmission of COVID-19. JAMA 2020;323(18):1837-8.
6. Brooks JT, Beezhold DH, Noti JD, et al. Maximizing Fit for Cloth and Medical Procedure Masks to Improve Performance and Reduce SARS-CoV-2 Transmission and Exposure, 2021. MMWR Morb Mortal Wkly Rep 2021;70(7):254-7.
7. Zhang X, Wang J. Dose-response Relation Deduced for Coronaviruses from COVID-19, SARS and MERS Meta-analysis Results and its Application for Infection Risk Assessment of Aerosol Transmission. Clin Infect Dis [Internet] 2020;Available from: http://dx.doi.org/10.1093/cid/ciaa1675
8. Hub SLK. The Logistics Challenges of COVID-19 Vaccination Distribution - Supply Chain 24/7 [Internet]. [cited 2021 Mar 8];Available from: https://www.supplychain247.com/article/the_logistics_challenges_of_covid_19_vaccination_distribution
9. Sah R, Tribhuvan University Teaching Hospital, Institute of Medicine, Kathmandu, Nepal, Roy N, et al. THE FIRST REPORT OF A POSSIBLE SARS-CoV-2 REINFECTION IN NEPAL. J exp biol agric sci 2021;9(1):1-4.
10. The New York Times. More Than One-Third of U.S. Coronavirus Deaths Are Linked to Nursing Homes [Internet]. The New York Times. 2021 [cited 2021 Mar 8];Available from: https://www.nytimes.com/interactive/2020/us/coronavirus-nursing-homes.html
11. Jefferson T, Del Mar CB, Dooley L, et al. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev 2011;(7):CD006207.
12. Oltermann P. Germany weighs up mandatory FFP2 masks in shops and on transport [Internet]. The Guardian. 2021 [cited 2021 Feb 25];Available from: http://www.theguardian.com/world/2021/jan/18/germany-weighs-up-mandatory-ffp2-masks-in-shops-and-on-transport

ELIGIBILITY:
Study inclusion criteria;

* Written informed consent
* Healthcare workers at nursing homes with resident contact
* Willingness to adhere to study protocol

Additional inclusion criteria for primary objective 2 (reinfection after vaccination)

- SARS-CoV-2 vaccination

List the study exclusion criteria:

* Unwillingness to adhere to study protocol
* HCW exclusively working with patients with aerosol-generating procedures during the entire study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-04-08 (Estimated); Primary Completion 2021-07-08 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | 16 weeks
  The primary endpoint is new SARS-CoV-2 infections among healthcare workers, measured by weekly, pooled saliva specimen-based SARS-CoV-2 testing.

SECONDARY OUTCOMES:
Exposure based on behavior | 16 weeks
  Secondary outcomes are questionnaires on monthly activity for healthcare workers; focus group discussions on workplace vs. private exposure to COVID-19 patients. All healthcare workers are tested by serology testing at baseline. Serology testing and saliva-based PCR-testing for healthcare workers are voluntary and are performed upon written informed consent.

CONTACTS AND LOCATIONS:
Locations (1):
- Gesundheitszentren für das Alter, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Nair S, Jones MA, Thorning S, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD006207. doi: 10.1002/14651858.CD006207.pub4. PMID 21735402
- [Background] Li P, Fu JB, Li KF, Liu JN, Wang HL, Liu LJ, Chen Y, Zhang YL, Liu SL, Tang A, Tong ZD, Yan JB. Transmission of COVID-19 in the terminal stages of the incubation period: A familial cluster. Int J Infect Dis. 2020 Jul;96:452-453. doi: 10.1016/j.ijid.2020.03.027. Epub 2020 Mar 16. PMID 32194239
- [Background] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Background] Cole EC, Cook CE. Characterization of infectious aerosols in health care facilities: an aid to effective engineering controls and preventive strategies. Am J Infect Control. 1998 Aug;26(4):453-64. doi: 10.1016/s0196-6553(98)70046-x. PMID 9721404
- [Background] Bourouiba L. Turbulent Gas Clouds and Respiratory Pathogen Emissions: Potential Implications for Reducing Transmission of COVID-19. JAMA. 2020 May 12;323(18):1837-1838. doi: 10.1001/jama.2020.4756. No abstract available. PMID 32215590
- [Background] Wei J, Li Y. Airborne spread of infectious agents in the indoor environment. Am J Infect Control. 2016 Sep 2;44(9 Suppl):S102-8. doi: 10.1016/j.ajic.2016.06.003. PMID 27590694
- [Background] Zhang X, Wang J. Dose-response Relation Deduced for Coronaviruses From Coronavirus Disease 2019, Severe Acute Respiratory Syndrome, and Middle East Respiratory Syndrome: Meta-analysis Results and its Application for Infection Risk Assessment of Aerosol Transmission. Clin Infect Dis. 2021 Jul 1;73(1):e241-e245. doi: 10.1093/cid/ciaa1675. PMID 33119733